CLINICAL TRIAL: NCT00414440
Title: A Multicenter, Randomized, Placebo-controlled, Double-blind Study on the Efficacy, Safety and Tolerability of Everolimus in Preventing End-stage Renal Disease (ESRD) in Patients With Autosomal Dominant Polycystic Kidney Disease (ADPKD)
Brief Title: Efficacy, Safety and Tolerability of Everolimus in Preventing End-stage Renal Disease in Patients With Autosomal Dominant Polycystic Kidney Disease
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CRAD001ADE12; 2006-001485-16
Record Dates: First submitted 2006-12-20; First posted 2006-12-21 (Estimated); Results first posted 2015-01-14 (Estimated); Last update posted 2015-01-14 (Estimated); Status verified 2015-01

CONDITIONS: Autosomal Dominant Polycystic Kidney Disease
Keywords: end-stage renal disease, ESRD, autosomal dominant polycystic kidney disease, ADPKD, everolimus
MeSH Terms: conditions — Polycystic Kidney, Autosomal Dominant; Kidney Failure, Chronic | interventions — Everolimus

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor

ARMS (2):
- Everolimus (Experimental): Patients in the everolimus group initially received 5 mg/day everolimus divided in 2 equal doses (i.e. 2.5 mg b.i.d.). Dose adjustments were performed to achieve a blood trough level of 3-8 ng/mL (maximum daily dose: 10 mg/day [5 mg b.i.d.]).
  Interventions: Drug: Everolimus
- Placebo (Placebo Comparator): Placebo tablets equivalent to the dosage of everolimus 5 mg/day, divided in 2 equal doses.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Placebo — placebo comparator
  Arms: Placebo
Drug: Everolimus — experimental
  Other Names: certican
  Arms: Everolimus

SUMMARY:
This study will assess whether everolimus (RAD001) is effective in preventing cyst and kidney expansion as well as worsening of renal function in patients with ADPKD and whether the application of 5 mg/day everolimus as monotherapy is safe and well tolerated.

ELIGIBILITY:
Inclusion Criteria

1. Clinical diagnosis of autosomal dominant polycystic kidney disease ADPKD
2. Chronic kidney disease (CKD) stage II / III
3. Females capable of becoming pregnant must have a negative serum pregnancy test within 7 days prior to or at baseline, and are required to practice an approved method of birth control for the duration of the study and for a period of 6 weeks following discontinuation of study medication, even where there has been a history of infertility

Exclusion Criteria

1. ADPKD patients with normal renal function
2. ADPKD patients with CKD stage IV
3. Patients with a history of subarachnoid bleeding
4. Patients with a history of severe infections
5. Patients with life-threatening urinary tract or cyst infection in the past
6. Patients who have received any investigational drug within four weeks prior to baseline
7. Patients who have been treated with any non-protocol immunosuppressive drug or treatment within one month prior to baseline

Other protocol-defined inclusion/exclusion criteria may apply

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 431 (Actual)
Dates: Start 2006-12; Primary Completion 2013-10 (Actual); Study Completion 2013-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (23):
- Austria (3):
  - Novartis Investigative Site, Innsbruck
  - Novartis Investigative Site, Linz
  - Novartis Investigative Site, Vienna
- France (5):
  - Novartis Investigative Site, Brest
  - Novartis Investigative Site, Grenoble
  - Novartis Investigative Site, Nantes
  - Novartis Investigative Site, Paris
  - Novartis Investigative Site, Toulouse
- Germany (15):
  - Novartis Investigative Site, Berlin
  - Novartis Investigative Site, Cologne
  - Novartis Investigative Site, Erlangen
  - Novartis Investigative Site, Essen
  - Novartis Investigative Site, Frankfurt am Main
  - Novartis Investigative Site, Freiburg im Breisgau
  - Novartis Investigative Site, Hamburg
  - Novartis Investigative Site, Heidelberg
  - Novartis Investigative Site, Homburg
  - Novartis Investigative Site, Kiel
  - Novartis Investigative Site, Leipzig
  - Novartis Investigative Site, Lübeck
  - Novartis Investigative Site, Münster
  - Novartis Investigative Site, Regensburg
  - Novartis Investigative Site, Würzburg

REFERENCES:
- [Derived] St Pierre K, Cashmore BA, Bolignano D, Zoccali C, Ruospo M, Craig JC, Strippoli GF, Mallett AJ, Green SC, Tunnicliffe DJ. Interventions for preventing the progression of autosomal dominant polycystic kidney disease. Cochrane Database Syst Rev. 2024 Oct 2;10(10):CD010294. doi: 10.1002/14651858.CD010294.pub3. PMID 39356039
- [Derived] Walz G, Budde K, Mannaa M, Nurnberger J, Wanner C, Sommerer C, Kunzendorf U, Banas B, Horl WH, Obermuller N, Arns W, Pavenstadt H, Gaedeke J, Buchert M, May C, Gschaidmeier H, Kramer S, Eckardt KU. Everolimus in patients with autosomal dominant polycystic kidney disease. N Engl J Med. 2010 Aug 26;363(9):830-40. doi: 10.1056/NEJMoa1003491. Epub 2010 Jun 26. PMID 20581392

RESULTS

PARTICIPANT FLOW:
Period: Core Period
Arm/Group | Everolimus | Placebo
Started | 214 (Core period) | 217 (Core period)
Completed | 144 (Core period) | 185 (Core period)
Not Completed | 70 | 32
Not completed — Withdrawal by Subject | 70 | 32
Period: Extension Period
Arm/Group | Everolimus | Placebo
Started | 214 (Extension) | 217 (Extension)
Completed | 64 (Extension) | 77 (Extension)
Not Completed | 150 | 140
Not completed — Lost to Follow-up | 44 | 52
Not completed — Did not consent to continue follow up | 61 | 54
Not completed — Other | 1 | 1
Not completed — Administrative | 16 | 16
Not completed — Death | 1 | 2
Not completed — Withdrawal by Subject | 9 | 7
Not completed — Not included in follow up period | 18 | 8

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Everolimus | Placebo | Total
Number analyzed (Participants) | 214 | 217 | 431
Age, Continuous [Mean (Standard Deviation); unit: years] — Average age of participants
  years | 44.6 (10.1) | 44.5 (10.4) | 44.5 (10.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 105 | 117 | 222
  Male | 109 | 100 | 209
Race/Ethnicity, Customized [Number; unit: participants]
  Asian Oriental | 4 | 0 | 4
  Black or African American | 1 | 0 | 1
  White | 208 | 217 | 425
  Other, Unknown or Not Reported | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Primary Efficacy Analysis of Total Kidney Volume (mITT Set, Multiple Imputation)
Description: Everolimus (RAD001) compared to placebo with respect to the change from baseline in total kidney volume at Month 24.
Time Frame: Baseline, Month 24
Population: mITT set
Measure: Mean (95% Confidence Interval); unit: mL
Arm/Group | Everolimus | Placebo
Number analyzed (Participants) | 214 | 217
mL | 230.1 [172.4 to 287.9] | 300.8 [247.5 to 354.1]

2. Secondary Outcome: Course of Calculated GFR (mL/Min/1.73 m^2) From Month 24 to Month 60
Description: Course of calculated GFR (mL/min/1.73 m^2) at Months 24, 36, 48 and 60
Time Frame: Months 24, 36, 48 and 60
Population: ITT
Measure: Mean (Standard Deviation); unit: mL/min/1.73 m^2
Arm/Group | Everolimus | Placebo
Number analyzed (Participants) | 214 | 217
mL/min/1.73 m^2
  Month 24 | 43.9 (23.9) | 48.8 (20.8)
  Month 36 | 42.6 (23.5) | 44.9 (22.2)
  Month 48 | 39.6 (22.2) | 42.7 (22.5)
  Month 60 | 37.7 (23.8) | 37.6 (21.6)

3. Secondary Outcome: Calculated GFR, Change From Baseline at Month 60 by Baseline cGFR
Description: Change in renal function was assessed by the estimated Glomerular Filtration Rate (eGFR) using the abbreviated (4 variables) Modification of Diet in Renal Disease (MDRD-4) formula which was developed by the MDRD Study Group and has been validated in patients with chronic kidney disease. The MDRD-4 formula used for the eGFR calculation is: eGFR (mL/min/1.73m^2) = 186.3*(C^-1.154)*(A^-0.203)*G*R, where C is the serum concentration of creatinine (mg/dL), A is age (years), G=0.742 when gender is female, otherwise G=1, R=1.21 when race is black, otherwise R=1. The changes in renal function were analyzed via analysis of covariance (ANCOVA) with treatment, pre-transplant hepatitis C virus status and randomization eGFR as covariates. Based on these ANCOVA analyses, the least-squares mean and standard errors of change were reported.
Time Frame: Months 24, 36, 48 and 60
Population: ITT
Measure: Mean (Standard Deviation); unit: mL/min/1.73 m^2
Arm/Group | Everolimus | Placebo
Number analyzed (Participants) | 64 | 75
mL/min/1.73 m^2
  >70 mL/min/1.73 m^2 n=11, 18 | -14.8 (22.7) | -20.5 (11.1)
  ≤70 mL/min/1.73 m^2 n=53, 57 | -16.1 (17.6) | -15.6 (15.2)
  >60 mL/min/1.73 m^2 n=21.26 | -17.0 (17.3) | -20.0 (13.6)
  ≤60 mL/min/1.73 m^2 n=43,49 | -15.3 (19.0) | -15.1 (14.7)
  >50 mL/min/1.73 m^2 n=36,39 | -19.0 (17.3) | -19.4 (12.6)
  ≤50 mL/min/1.73 m^2 n=28, 36 | -11.8 (19.2) | -14.0 (15.8)

4. Secondary Outcome: Changes in Systolic Blood Pressure (SBP) and Diastolic Blood Pressure (DBP)
Description: Changes in systolic blood pressure (SBP) and diastolic blood pressure (DBP), at baseline and then months 12 and 24
Time Frame: Baseline, Months 12 and 24
Population: ITT, observed cases
Measure: Mean (Standard Deviation); unit: mmHG
Units Other Than Participants: mean
Arm/Group | Everolimus | Placebo
Number analyzed (Participants) | 213 | 216
Number analyzed (mean) | 213 | 216
mmHG
  Baseline SBP | 136 (16) | 135 (17)
  Month 12 SBP | 134 (15) | 134 (16)
  Month 24 SBP | 134 (17) | 134 (15)
  Baseline DBP | 88 (11) | 88 (10)
  Month 12 DBP | 86 (10) | 86 (10)
  Month 24 DBP | 85 (10) | 85 (10)

5. Secondary Outcome: Calculated GFR (mL/Min/1.73 m^2), Change From Baseline by Visit
Description: Change in renal function was assessed by the Glomerular Filtration Rate (GFR) using the abbreviated (4 variables) Modification of Diet in Renal Disease (MDRD-4) formula which was developed by the MDRD Study Group and has been validated in patients with chronic kidney disease. The MDRD-4 formula used for the eGFR calculation is: eGFR (mL/min/1.73m^2) = 186.3*(C^-1.154)*(A^-0.203)*G*R, where C is the serum concentration of creatinine (mg/dL), A is age (years), G=0.742 when gender is female, otherwise G=1, R=1.21 when race is black, otherwise R=1. The changes in renal function were analyzed via analysis of covariance (ANCOVA) with treatment, pre-transplant hepatitis C virus status and randomization eGFR as covariates. Based on these ANCOVA analyses, the least-squares mean and standard errors of change were reported.
Time Frame: Months 3, 6, 9, 12, 18 and 24
Population: ITT set, observed cases
Measure: Mean (Standard Deviation); unit: mL/min/1.73m^2
Units Other Than Participants: calculated GFR
Arm/Group | Everolimus | Placebo
Number analyzed (Participants) | 213 | 216
Number analyzed (calculated GFR) | 213 | 216
mL/min/1.73m^2
  Week 1 | 2.0 (5.9) | -0.9 (6.1)
  Week 2 | 1.7 (5.9) | -0.9 (6.5)
  Week 4 | 0.6 (6.3) | -1.2 (6.7)
  Month 3 | -0.5 (8.2) | -2.4 (6.7)
  Month 6 | -2.3 (7.7) | -2.2 (6.7)
  Month 9 | -4.6 (8.2) | -2.4 (6.0)
  Month 12 | -5.4 (7.5) | -3.2 (6.9)
  Month 18 | -7.7 (8.5) | -5.5 (6.7)
  Month 24 | -8.9 (8.8) | -7.7 (6.6)

ADVERSE EVENTS:
Arm/Group | Everolimus | Placebo
Serious Adverse Events (participants affected / at risk) | 80/214 | 51/217
Other Adverse Events (participants affected / at risk) | 205/214 | 185/217
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Everolimus (N=214) | Placebo (N=217)
ANAEMIA (Blood and lymphatic system disorders) | 2 | 0
IRON DEFICIENCY ANAEMIA (Blood and lymphatic system disorders) | 1 | 0
LEUKOCYTOSIS (Blood and lymphatic system disorders) | 1 | 0
LYMPH NODE PAIN (Blood and lymphatic system disorders) | 1 | 0
LYMPHADENOPATHY (Blood and lymphatic system disorders) | 1 | 0
NEUTROPENIA (Blood and lymphatic system disorders) | 1 | 0
ANGINA PECTORIS (Cardiac disorders) | 0 | 1
ATRIAL FIBRILLATION (Cardiac disorders) | 2 | 0
ATRIAL FLUTTER (Cardiac disorders) | 1 | 0
BRADYARRHYTHMIA (Cardiac disorders) | 0 | 1
BRADYCARDIA (Cardiac disorders) | 1 | 0
CARDIAC FAILURE (Cardiac disorders) | 1 | 0
CARDIOGENIC SHOCK (Cardiac disorders) | 1 | 0
CORONARY ARTERY DISEASE (Cardiac disorders) | 0 | 3
LEFT VENTRICULAR FAILURE (Cardiac disorders) | 1 | 0
MITRAL VALVE INCOMPETENCE (Cardiac disorders) | 1 | 0
MYOPERICARDITIS (Cardiac disorders) | 1 | 0
PERICARDIAL EFFUSION (Cardiac disorders) | 2 | 0
POLYCYSTIC LIVER DISEASE (Congenital, familial and genetic disorders) | 0 | 1
ACUTE VESTIBULAR SYNDROME (Ear and labyrinth disorders) | 0 | 1
VERTIGO (Ear and labyrinth disorders) | 0 | 1
GOITRE (Endocrine disorders) | 0 | 1
RETINAL DETACHMENT (Eye disorders) | 1 | 0
ABDOMINAL PAIN (Gastrointestinal disorders) | 2 | 1
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 2 | 1
ABDOMINAL TENDERNESS (Gastrointestinal disorders) | 1 | 0
APHTHOUS STOMATITIS (Gastrointestinal disorders) | 2 | 0
ASCITES (Gastrointestinal disorders) | 1 | 0
COLITIS (Gastrointestinal disorders) | 0 | 1
COLONIC POLYP (Gastrointestinal disorders) | 1 | 0
CROHN'S DISEASE (Gastrointestinal disorders) | 0 | 1
DIARRHOEA (Gastrointestinal disorders) | 3 | 1
GASTRIC HAEMORRHAGE (Gastrointestinal disorders) | 1 | 0
GASTRITIS (Gastrointestinal disorders) | 1 | 0
GASTRODUODENITIS (Gastrointestinal disorders) | 0 | 1
HAEMORRHOIDAL HAEMORRHAGE (Gastrointestinal disorders) | 1 | 0
INGUINAL HERNIA (Gastrointestinal disorders) | 2 | 4
OESOPHAGITIS (Gastrointestinal disorders) | 1 | 0
RECTAL HAEMORRHAGE (Gastrointestinal disorders) | 1 | 0
SUBILEUS (Gastrointestinal disorders) | 1 | 0
UMBILICAL HERNIA (Gastrointestinal disorders) | 3 | 2
VOMITING (Gastrointestinal disorders) | 1 | 0
ASTHENIA (General disorders) | 2 | 2
BLOODY DISCHARGE (General disorders) | 0 | 1
CHEST PAIN (General disorders) | 1 | 1
DISEASE PROGRESSION (General disorders) | 4 | 2
DRUG WITHDRAWAL SYNDROME (General disorders) | 0 | 1
OEDEMA (General disorders) | 1 | 0
OEDEMA PERIPHERAL (General disorders) | 1 | 0
PYREXIA (General disorders) | 1 | 1
CHOLECYSTITIS (Hepatobiliary disorders) | 1 | 0
HEPATIC CYST (Hepatobiliary disorders) | 1 | 1
HEPATIC CYST RUPTURED (Hepatobiliary disorders) | 1 | 1
HEPATOMEGALY (Hepatobiliary disorders) | 1 | 0
PORTAL VEIN THROMBOSIS (Hepatobiliary disorders) | 1 | 0
ANAPHYLACTIC SHOCK (Immune system disorders) | 1 | 0
HOUSE DUST ALLERGY (Immune system disorders) | 1 | 0
HYPERSENSITIVITY (Immune system disorders) | 1 | 0
ACUTE TONSILLITIS (Infections and infestations) | 1 | 0
ANOGENITAL WARTS (Infections and infestations) | 0 | 1
APPENDICITIS (Infections and infestations) | 1 | 0
BRONCHITIS (Infections and infestations) | 1 | 0
DIVERTICULITIS (Infections and infestations) | 0 | 1
ENTEROCOLITIS INFECTIOUS (Infections and infestations) | 1 | 0
ERYSIPELAS (Infections and infestations) | 0 | 1
GASTROENTERITIS (Infections and infestations) | 3 | 0
GASTROINTESTINAL INFECTION (Infections and infestations) | 1 | 1
HEPATIC CYST INFECTION (Infections and infestations) | 0 | 1
HERPES SIMPLEX (Infections and infestations) | 1 | 0
HERPES ZOSTER (Infections and infestations) | 2 | 0
HERPES ZOSTER OPHTHALMIC (Infections and infestations) | 1 | 0
INFECTION (Infections and infestations) | 2 | 0
INFECTIVE EXACERBATION OF CHRONIC OBSTRUCTIVE AIRWAYS DISEASE (Infections and infestations) | 0 | 1
LYMPH NODE TUBERCULOSIS (Infections and infestations) | 1 | 0
LYMPHADENITIS BACTERIAL (Infections and infestations) | 1 | 0
OTITIS MEDIA CHRONIC (Infections and infestations) | 1 | 0
PAPILLOMA VIRAL INFECTION (Infections and infestations) | 0 | 1
PNEUMONIA (Infections and infestations) | 5 | 1
PYELONEPHRITIS (Infections and infestations) | 1 | 2
PYELONEPHRITIS ACUTE (Infections and infestations) | 0 | 1
RENAL CYST INFECTION (Infections and infestations) | 2 | 4
RESPIRATORY TRACT INFECTION (Infections and infestations) | 0 | 2
SINUSITIS (Infections and infestations) | 2 | 0
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 1 | 1
UROSEPSIS (Infections and infestations) | 1 | 0
VESTIBULAR NEURONITIS (Infections and infestations) | 1 | 0
VIRAL INFECTION (Infections and infestations) | 0 | 1
ARTHROPOD STING (Injury, poisoning and procedural complications) | 1 | 0
CONJUNCTIVAL ABRASION (Injury, poisoning and procedural complications) | 0 | 1
CORNEAL ABRASION (Injury, poisoning and procedural complications) | 0 | 1
FOOT FRACTURE (Injury, poisoning and procedural complications) | 1 | 0
FOREIGN BODY IN EYE (Injury, poisoning and procedural complications) | 0 | 1
INCISIONAL HERNIA (Injury, poisoning and procedural complications) | 0 | 2
LIGAMENT INJURY (Injury, poisoning and procedural complications) | 0 | 1
MENISCUS LESION (Injury, poisoning and procedural complications) | 0 | 1
POST PROCEDURAL HAEMORRHAGE (Injury, poisoning and procedural complications) | 1 | 0
STERNAL FRACTURE (Injury, poisoning and procedural complications) | 0 | 1
BLOOD CREATINE PHOSPHOKINASE INCREASED (Investigations) | 1 | 1
BLOOD CREATININE INCREASED (Investigations) | 2 | 0
C-REACTIVE PROTEIN INCREASED (Investigations) | 3 | 0
WEIGHT DECREASED (Investigations) | 4 | 0
DIABETES MELLITUS (Metabolism and nutrition disorders) | 1 | 0
GOUT (Metabolism and nutrition disorders) | 1 | 0
HYPOKALAEMIA (Metabolism and nutrition disorders) | 1 | 0
ANKYLOSING SPONDYLITIS (Musculoskeletal and connective tissue disorders) | 0 | 1
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 2 | 0
ARTHRITIS REACTIVE (Musculoskeletal and connective tissue disorders) | 1 | 0
BACK PAIN (Musculoskeletal and connective tissue disorders) | 1 | 0
FLANK PAIN (Musculoskeletal and connective tissue disorders) | 2 | 1
FOOT DEFORMITY (Musculoskeletal and connective tissue disorders) | 1 | 0
INTERVERTEBRAL DISC PROTRUSION (Musculoskeletal and connective tissue disorders) | 1 | 0
MUSCULAR WEAKNESS (Musculoskeletal and connective tissue disorders) | 1 | 0
MYALGIA (Musculoskeletal and connective tissue disorders) | 4 | 1
MYOSITIS (Musculoskeletal and connective tissue disorders) | 1 | 0
POLYARTHRITIS (Musculoskeletal and connective tissue disorders) | 1 | 0
RHABDOMYOLYSIS (Musculoskeletal and connective tissue disorders) | 1 | 1
ADENOCARCINOMA PANCREAS (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
BENIGN OVARIAN TUMOUR (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
BREAST CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
CHOLESTEATOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
PANCREATIC CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
PLASMACYTOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
THYROID NEOPLASM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
UTERINE LEIOMYOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
CEREBRAL ATROPHY (Nervous system disorders) | 1 | 0
CEREBRAL HAEMORRHAGE (Nervous system disorders) | 1 | 0
CEREBROVASCULAR ACCIDENT (Nervous system disorders) | 1 | 1
HEMIPARESIS (Nervous system disorders) | 0 | 1
MIGRAINE (Nervous system disorders) | 0 | 1
MIGRAINE WITH AURA (Nervous system disorders) | 0 | 1
NEUROPATHY PERIPHERAL (Nervous system disorders) | 0 | 1
RUPTURED CEREBRAL ANEURYSM (Nervous system disorders) | 1 | 0
SYNCOPE (Nervous system disorders) | 0 | 2
PREGNANCY (Pregnancy, puerperium and perinatal conditions) | 1 | 0
ACUTE PSYCHOSIS (Psychiatric disorders) | 1 | 0
DEPRESSED MOOD (Psychiatric disorders) | 1 | 0
DEPRESSION (Psychiatric disorders) | 1 | 1
PARANOIA (Psychiatric disorders) | 1 | 0
PSYCHOTIC DISORDER (Psychiatric disorders) | 0 | 1
SUICIDE ATTEMPT (Psychiatric disorders) | 1 | 0
CALCULUS URETERIC (Renal and urinary disorders) | 1 | 0
HAEMATURIA (Renal and urinary disorders) | 2 | 0
NEPHROTIC SYNDROME (Renal and urinary disorders) | 1 | 0
RENAL COLIC (Renal and urinary disorders) | 2 | 1
RENAL CYST RUPTURED (Renal and urinary disorders) | 0 | 1
RENAL FAILURE (Renal and urinary disorders) | 1 | 0
RENAL FAILURE ACUTE (Renal and urinary disorders) | 5 | 1
RENAL HAEMORRHAGE (Renal and urinary disorders) | 3 | 2
RENAL IMPAIRMENT (Renal and urinary disorders) | 2 | 1
BREAST DISCHARGE (Reproductive system and breast disorders) | 0 | 1
BREAST FIBROSIS (Reproductive system and breast disorders) | 0 | 1
BREAST HYPERPLASIA (Reproductive system and breast disorders) | 0 | 1
COLPOCELE (Reproductive system and breast disorders) | 0 | 1
DYSMENORRHOEA (Reproductive system and breast disorders) | 1 | 0
MENORRHAGIA (Reproductive system and breast disorders) | 1 | 0
MENSTRUATION IRREGULAR (Reproductive system and breast disorders) | 1 | 0
OVARIAN CYST (Reproductive system and breast disorders) | 7 | 0
PELVIC FLUID COLLECTION (Reproductive system and breast disorders) | 1 | 0
POLYCYSTIC OVARIES (Reproductive system and breast disorders) | 1 | 0
VAGINAL HAEMORRHAGE (Reproductive system and breast disorders) | 2 | 0
CHRONIC OBSTRUCTIVE PULMONARY DISEASE (Respiratory, thoracic and mediastinal disorders) | 1 | 0
COUGH (Respiratory, thoracic and mediastinal disorders) | 1 | 1
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 1 | 0
DYSPNOEA EXERTIONAL (Respiratory, thoracic and mediastinal disorders) | 1 | 0
LUNG DISORDER (Respiratory, thoracic and mediastinal disorders) | 1 | 0
PAINFUL RESPIRATION (Respiratory, thoracic and mediastinal disorders) | 1 | 0
PLEURAL EFFUSION (Respiratory, thoracic and mediastinal disorders) | 1 | 0
PLEURISY (Respiratory, thoracic and mediastinal disorders) | 1 | 0
PNEUMONITIS (Respiratory, thoracic and mediastinal disorders) | 2 | 0
PULMONARY EMBOLISM (Respiratory, thoracic and mediastinal disorders) | 0 | 1
PULMONARY OEDEMA (Respiratory, thoracic and mediastinal disorders) | 1 | 0
ANGIOEDEMA (Skin and subcutaneous tissue disorders) | 8 | 0
HYPOAESTHESIA FACIAL (Skin and subcutaneous tissue disorders) | 0 | 1
ANGIODYSPLASIA (Vascular disorders) | 1 | 0
DEEP VEIN THROMBOSIS (Vascular disorders) | 0 | 2
HYPERTENSION (Vascular disorders) | 0 | 1
HYPERTENSIVE CRISIS (Vascular disorders) | 0 | 1
HYPOTENSION (Vascular disorders) | 1 | 0
ILIAC ARTERY STENOSIS (Vascular disorders) | 0 | 1
INTERMITTENT CLAUDICATION (Vascular disorders) | 0 | 1
PERIPHERAL ARTERIAL OCCLUSIVE DISEASE (Vascular disorders) | 0 | 1
THROMBOSIS (Vascular disorders) | 1 | 0
VARICOSE VEIN (Vascular disorders) | 0 | 1
VASCULITIS (Vascular disorders) | 0 | 1
VENOUS THROMBOSIS LIMB (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Everolimus (N=214) | Placebo (N=217)
ANAEMIA (Blood and lymphatic system disorders) | 35 | 11
LEUKOPENIA (Blood and lymphatic system disorders) | 38 | 6
THROMBOCYTOPENIA (Blood and lymphatic system disorders) | 30 | 2
ABDOMINAL DISCOMFORT (Gastrointestinal disorders) | 12 | 8
ABDOMINAL PAIN (Gastrointestinal disorders) | 24 | 13
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 14 | 13
APHTHOUS STOMATITIS (Gastrointestinal disorders) | 83 | 12
DIARRHOEA (Gastrointestinal disorders) | 48 | 34
NAUSEA (Gastrointestinal disorders) | 20 | 12
VOMITING (Gastrointestinal disorders) | 11 | 14
ASTHENIA (General disorders) | 11 | 6
FATIGUE (General disorders) | 20 | 19
OEDEMA (General disorders) | 25 | 12
OEDEMA PERIPHERAL (General disorders) | 42 | 20
PYREXIA (General disorders) | 12 | 9
BRONCHITIS (Infections and infestations) | 21 | 23
GASTROENTERITIS (Infections and infestations) | 11 | 4
NASOPHARYNGITIS (Infections and infestations) | 83 | 83
ORAL HERPES (Infections and infestations) | 15 | 4
SINUSITIS (Infections and infestations) | 14 | 13
URINARY TRACT INFECTION (Infections and infestations) | 22 | 19
BLOOD CREATINE PHOSPHOKINASE INCREASED (Investigations) | 32 | 15
BLOOD CREATININE INCREASED (Investigations) | 38 | 13
HYPERCHOLESTEROLAEMIA (Metabolism and nutrition disorders) | 46 | 8
HYPERLIPIDAEMIA (Metabolism and nutrition disorders) | 28 | 5
HYPERTRIGLYCERIDAEMIA (Metabolism and nutrition disorders) | 15 | 8
HYPERURICAEMIA (Metabolism and nutrition disorders) | 7 | 13
IRON DEFICIENCY (Metabolism and nutrition disorders) | 12 | 2
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 13 | 5
BACK PAIN (Musculoskeletal and connective tissue disorders) | 15 | 17
FLANK PAIN (Musculoskeletal and connective tissue disorders) | 17 | 23
MUSCLE SPASMS (Musculoskeletal and connective tissue disorders) | 10 | 12
MYALGIA (Musculoskeletal and connective tissue disorders) | 14 | 3
HEADACHE (Nervous system disorders) | 37 | 27
HAEMATURIA (Renal and urinary disorders) | 13 | 9
PROTEINURIA (Renal and urinary disorders) | 28 | 15
COUGH (Respiratory, thoracic and mediastinal disorders) | 24 | 19
OROPHARYNGEAL PAIN (Respiratory, thoracic and mediastinal disorders) | 12 | 9
ACNE (Skin and subcutaneous tissue disorders) | 30 | 6
RASH (Skin and subcutaneous tissue disorders) | 18 | 8
HYPERTENSION (Vascular disorders) | 33 | 29

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Other disclosure agreement that restricts the right of the PI to discuss or publish trial results after the trial is completed.

The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial; or disclosure of the trial results in their entirety.